CLINICAL TRIAL: NCT05724849
Title: Venlafaxine for the Prevention of Depression in Patients With Head and Neck Cancer
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: Issues with funding
Sponsor: Vanderbilt University Medical Center (Other)
Responsible Party: Principal Investigator, Michael Topf, Assistant Professor, Department of Otolaryngology, Vanderbilt University Medical Center
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: 230054
Record Dates: First submitted 2023-01-31; First posted 2023-02-13 (Actual); Last update posted 2024-01-18 (Actual); Status verified 2024-01

CONDITIONS: Head and Neck Cancer; Depression
MeSH Terms: conditions — Head and Neck Neoplasms; Depression | interventions — Venlafaxine Hydrochloride

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (3):
- Venlafaxine (Experimental): Patients who screen negative or meet criteria for mild MDD are eligible for the randomized control trial (RCT) portion of this study in which patients are randomized into either the intervention (venlafaxine) arm or placebo. Participants randomized into the intervention group will be prescribed a starting dose of venlafaxine immediate release (IR) 75mg once daily. The dosing will be increased at the following rate:
  Week 1: 75mg in AM
  Week 2: 75mg BID
  Week 3: 150mg in AM, 75mg in PM
  Week 4: 150mg BID
  For patients with hepatic impairment, severe renal impairment, or end stage kidney disease, the starting dose is 37.5 mg once daily, increased by increments of 37.5 mg per day to reach a maximum of 187.5 mg per day, given in two divided doses.
  Interventions: Drug: Venlafaxine
- Placebo (Placebo Comparator): Patients who screen negative or meet criteria for mild MDD are eligible for the randomized control trial (RCT) portion of this study in which patients are randomized into either the intervention (venlafaxine) arm or placebo. Participants randomized to the placebo group will receive a placebo capsule with the same dosing schedule as the intervention group.
  Interventions: Drug: Placebo
- Observation (Other): Patients who screen positive for moderate, moderately-severe, or severe MDD are excluded from the RCT and will be enrolled in the study as an observation cohort. These patients will be offered initiation of venlafaxine and will be referred to our collaborating oncologic psychiatrist. Patients in cohort B will still complete the same patient-reported outcome measures (PROMs) as patients in cohort A, allowing us to collect data and better understand what effects venlafaxine has on patients who are already diagnosed with depression at the start of treatment for HNC.
  Interventions: Drug: Venlafaxine

INTERVENTIONS:
Drug: Venlafaxine — See arm/group description.
  Other Names: Effexor
  Arms: Observation; Venlafaxine
Drug: Placebo — See arm/group description.
  Arms: Placebo

SUMMARY:
This is a pilot double-blinded, randomized, placebo-controlled trial to determine if venlafaxine prevents depression in patients undergoing surgery for Head and Neck Cancer (HNC).

DETAILED DESCRIPTION:
Patients with head and neck cancer (HNC) are disproportionately affected by major depressive disorder (MDD), with up to 50% developing MDD compared to 15-25% of patients with other solid malignancies. The higher rates of depression seen in HNC patients are likely related to treatment-associated disfigurement, voice and swallow dysfunction, and other physical alterations that significantly diminish quality of life. Survivors of HNC have a significantly increased risk of suicide when compared to other cancers. The rate of suicide among HNC survivors is 63.4 suicides per 100,000 person-years, which is three times that of other cancer survivors and second highest only behind pancreatic cancer.

There is evidence to suggest that depression plays a role in HNC prognosis, with studies showing a 25% decrease in overall survival in HNC patients with depression. Despite the prevalence and impact of depression in HNC patients, there has only been one randomized control trial to prevent depression in patients with HNC that showed potential benefit. This study used escitalopram, a selective-serotonin reuptake inhibitor (SSRI). A more appropriate medication would be one that provided mood stabilization as well as pain modulation, since it is known that HNC treatment can lead to long-term opioid use. Serotonin-norepinephrine reuptake inhibitors (SNRIs) provide dual action against serotonergic and noradrenergic receptors and have shown to provide superior pain relief than monoaminergic drugs such as SSRIs.

The investigators hypothesize that venlafaxine will provide mood stabilization and improved pain control in patients undergoing surgical treatment for HNC. The investigators plan to conduct a pilot double-blinded, randomized, placebo-controlled trial using venlafaxine in HNC patients treated with surgery. Patients who screen negative for Bipolar disorder (BPD) based on the screening tool The Mood Disorder Questionnaire (MDQ) as well as for MDD using the Patient Health Questionnaire (PHQ-9) preoperatively (Cohort A) will be randomized to either venlafaxine or placebo and will be assessed throughout the perioperative period with a series of validated self-reported questionnaires regarding depression, anxiety, pain, and other quality of life measures.

ELIGIBILITY:
Inclusion Criteria:

COHORT A (RCT)

1. Provision of signed and dated informed consent form
2. Stated willingness to comply with all study procedures and availability for the duration of the study
3. Male or female, aged 18 years or older
4. Have a recently diagnosed cutaneous or mucosal malignancy
5. Scheduled to undergo surgical treatment for their malignancy with curative intent
6. Ability to take medication orally or via gastric tube feeds
7. Willing to adhere to the study drug's dosing protocol
8. Score <10 on the PHQ-9

COHORT B (Observation cohort)

1. Provision of signed and dated informed consent form
2. Stated willingness to comply with all study procedures and availability for the duration of the study
3. Male or female, aged 18 years or older
4. Have a recently diagnosed cutaneous or mucosal malignancy
5. Scheduled to undergo surgical treatment for their malignancy with curative intent
6. Ability to take medication orally or via gastric tube feeds
7. Willing to adhere to the study drug's dosing protocol
8. Score >10 on the PHQ-9

Exclusion Criteria:

COHORT A (RCT)

1. Score >10 on PHQ-9
2. Score between 5-9 on PHQ-9 and elect for psychotherapy
3. Age less than 18 years
4. Primary malignancy of thyroid or parathyroid origin
5. Currently meet diagnostic criteria for psychosis, schizophrenia, or bipolar disorder
6. Currently receiving medication as treatment for depression or anxiety including: MAO inhibitors, Linezolid, Other SNRIs or SSRIs, Bupropion
7. Known allergic reaction to components of study drug
8. Treatment with another investigational drug or other intervention within 30 days
9. Females of child-bearing age who are pregnant or nursing
10. Inability to speak or understand English

COHORT B (Observation cohort)

1. Score <10 on PHQ-9
2. Unwillingness or inability to take venlafaxine
3. Age less than 18 years
4. Primary malignancy of thyroid or parathyroid origin
5. Currently receiving medication as treatment for depression or anxiety including: MAO inhibitors, Linezolid, Other SNRIs or SSRIs, Bupropion

7. Known allergic reaction to components of study drug 8. Treatment with another investigational drug or other intervention within 30 days 9. Females of child-bearing age who are pregnant or nursing 10. Inability to speak or understand English

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2023-08-01 (Estimated); Primary Completion 2026-08-01 (Estimated); Study Completion 2026-08-01 (Estimated)

PRIMARY OUTCOMES:
Prevention of Depression | 4 months post-operatively
  Rate of depression at any time interval within the 4-month post-surgery period in patients with no or mild MDD. This will be assessed using the Patient-Health Questionnaire (PHQ-9) which is scored ranging from 0-27 with a higher score indicating more severe depression. Four months was chosen as the duration to capture the adjuvant radiation period, which is typically 3 months post-surgery.

SECONDARY OUTCOMES:
Treatment of Depression | 4 months post-operatively
  Rate of depression at 4 months post-surgery in patients who initially screened positive for moderate, moderately-severe, or severe MDD. This will be assessed using the Patient-Health Questionnaire (PHQ-9) which is scored ranging from 0-27 with a higher score indicating more severe depression.
Prevention of Anxiety | 4 months post-operatively
  Rate of anxiety at 4-months post-surgery in all patients enrolled. This will be assessed using the Generalized Anxiety Disorder-7 (GAD-7) which reports scores on a scale, ranging from 0 to 21 with higher scores indicating worse outcomes.
Prevention of Pain | 4 months post-operatively
  Rate of pain control at 4-months post-surgery in all patients enrolled. This will be assessed using the Brief Pain Inventory-short form which is scored on a scale of 0 to 10 with a higher score indicating a worse outcome.
Prevention of Pain | 4 months post-operatively
  Duration of opioid use post-surgery in all patients enrolled. This will be assessed using the opioid diary.
Quality of Life Improvement | 4 months post-operatively
  Quality of life at 4 months post-surgery in all patients enrolled. This will be assessed using the FACE-Q HNC which is scored on a scale. The scale ranges from 0 to 100 with a higher score meaning a better outcome.

CONTACTS AND LOCATIONS:
Overall Officials: Michael C Topf, MD, Principal Investigator — Vanderbilt University Medical Center

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Lydiatt WM, Moran J, Burke WJ. A review of depression in the head and neck cancer patient. Clin Adv Hematol Oncol. 2009 Jun;7(6):397-403. PMID 19606075
- [Background] Chhabria KS, Carnaby GD. Psychometric validation of the Center for Epidemiological Studies Depression Scale in Head and Neck Cancer patients. Oral Oncol. 2017 Dec;75:158-162. doi: 10.1016/j.oraloncology.2017.11.010. Epub 2017 Nov 15. PMID 29224813
- [Background] Rieke K, Schmid KK, Lydiatt W, Houfek J, Boilesen E, Watanabe-Galloway S. Depression and survival in head and neck cancer patients. Oral Oncol. 2017 Feb;65:76-82. doi: 10.1016/j.oraloncology.2016.12.014. Epub 2017 Jan 1. PMID 28109472
- [Background] Archer J, Hutchison I, Korszun A. Mood and malignancy: head and neck cancer and depression. J Oral Pathol Med. 2008 May;37(5):255-70. doi: 10.1111/j.1600-0714.2008.00635.x. Epub 2008 Feb 26. PMID 18312300
- [Background] Cramer JD, Johnson JT, Nilsen ML. Pain in Head and Neck Cancer Survivors: Prevalence, Predictors, and Quality-of-Life Impact. Otolaryngol Head Neck Surg. 2018 Nov;159(5):853-858. doi: 10.1177/0194599818783964. Epub 2018 Jun 26. PMID 29943677
- [Background] Friedland CJ. Head and Neck Cancer: Identifying Depression as a Comorbidity Among Patients. Clin J Oncol Nurs. 2019 Feb 1;23(1):99-102. doi: 10.1188/19.CJON.99-102. PMID 30681992
- [Background] Barber B, Dergousoff J, Slater L, Harris J, O'Connell D, El-Hakim H, Biron VL, Mitchell N, Seikaly H. Depression and Survival in Patients With Head and Neck Cancer: A Systematic Review. JAMA Otolaryngol Head Neck Surg. 2016 Mar;142(3):284-8. doi: 10.1001/jamaoto.2015.3171. PMID 26796781
- [Background] Lydiatt WM, Denman D, McNeilly DP, Puumula SE, Burke WJ. A randomized, placebo-controlled trial of citalopram for the prevention of major depression during treatment for head and neck cancer. Arch Otolaryngol Head Neck Surg. 2008 May;134(5):528-35. doi: 10.1001/archotol.134.5.528. PMID 18490576
- [Background] Lydiatt WM, Bessette D, Schmid KK, Sayles H, Burke WJ. Prevention of depression with escitalopram in patients undergoing treatment for head and neck cancer: randomized, double-blind, placebo-controlled clinical trial. JAMA Otolaryngol Head Neck Surg. 2013 Jul;139(7):678-86. doi: 10.1001/jamaoto.2013.3371. PMID 23788218
- [Background] Panwar A, Rieke K, Burke WJ, Sayles H, Lydiatt WM; Prevention of Depression in Patients Being Treated for Head and Neck Cancer Trial (PROTECT) study group. Identification of Baseline Characteristics Associated With Development of Depression Among Patients With Head and Neck Cancer: A Secondary Analysis of a Randomized Clinical Trial. JAMA Otolaryngol Head Neck Surg. 2018 Nov 1;144(11):1004-1010. doi: 10.1001/jamaoto.2018.2228. PMID 30286230
- [Background] Smith EM, Pang H, Cirrincione C, Fleishman S, Paskett ED, Ahles T, Bressler LR, Fadul CE, Knox C, Le-Lindqwister N, Gilman PB, Shapiro CL; Alliance for Clinical Trials in Oncology. Effect of duloxetine on pain, function, and quality of life among patients with chemotherapy-induced painful peripheral neuropathy: a randomized clinical trial. JAMA. 2013 Apr 3;309(13):1359-67. doi: 10.1001/jama.2013.2813. PMID 23549581